CLINICAL TRIAL: NCT01481038
Title: Anticipative Diagnosis of Central Venous Catheter Related Bloodstream Infections Using Biphasic PNA FISH and Gram Stain/AOLC Tests
Brief Title: Anticipative Diagnosis of Central Venous Catheter Related Bloodstream Infections
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Robert Krause, MD, Univ.Prof.Dr, Medical University of Graz
Other Study IDs: CRBSI FFG Bridge
Record Dates: First submitted 2011-11-16; First posted 2011-11-29 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-05

CONDITIONS: Bloodstream Infection Due to Central Venous Catheter
Keywords: early detection; CRBSI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group dialysis patients: Patient on hemodialysis with central venous catheter
- Group hematology patients: Patients with hemato-oncologic underlying disease (plus/minus hematopoietic stem cell transplantation HSCT) and central venous catheter

SUMMARY:
Up to date methods for diagnosis of Catheter Related Bloodstream Infections (CRBSI) are performed only when CRBSI is clinically suspected. Thus, patients may actually suffer from CRBSI and are at risk to concurrently suffer from or develop complications like endocarditis or septic embolism when diagnostic procedures for the detection of CRBSI are introduced. The aim of the project is to investigate a more sensitive and specific test for anticipative diagnosis of CRBSI using biphasic PNA FISH test compared to Gram stain/AOLC test.

DETAILED DESCRIPTION:
Management of patients with hematologic malignancies, renal failure or diseases requiring intensive care often necessitates the use of central venous catheters (CVC). Beside obvious advantages CVCs bear a great risk for local or systemic infections. In the US estimated 250 000 catheter-related blood stream infection (CRBSIs) occur each year with mortality rates of 12-25%. Diagnosis of CRBSIs remains challenging as systemic clinical signs are unspecific and local signs of infection are often absent. Conventional methods for diagnosing CRBSIs require removal of the CVC. However, only 15% of CVCs removed in patients with clinical suspicion of CRBSI prove to be infected. It has been shown that CRBSI can also be detected by the differential time to positivity (DTP) method without catheter removal. The Gram stain/acridine-orange leukocyte cytospin (AOLC) test and PNA FISH test are another methods for the diagnosis of CRBSI that does not require the removal of the CVC and additionally have shown to be fast. Up to date methods for diagnosis of CRBSI are performed only when CRBSI is clinically suspected. Thus, patients may actually suffer from CRBSI and are at risk to concurrently suffer from or develop complications like endocarditis or septic embolism when diagnostic procedures for the detection of CRBSI are introduced. Since CRBSIs are not entirely preventable by strict hygiene measures earlier diagnosis of CRBSI in subclinical stages is desirable to avoid CRBSI-associated morbidity and mortality. Previously a pilot study showed that Gram stain/AOLC screening of CVCs in neutropenic patients was a useful test to predict the development of CRBSI on average 48 hours before the diagnosis was established by routine measures. In the pilot study Gram stain/AOLC screening test exhibited high specificity whereas sensitivity was moderate. PNA FISH is a specific slide-based staining technique that provides pathogen identification from blood samples containing a given amount of bacteria or fungi within a 1,5 hours. PNA FISH test has a slightly lower detection limit compared to Gram stain/AOLC which might therefore result in higher sensitivity when used as a screening tool. The aim of the project is to investigate a more sensitive and specific test for anticipative diagnosis of CRBSI using biphasic PNA FISH test compared to Gram stain/AOLC test.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing hemodialysis using a central venous catheter and
* Patients with underlying hematooncologic disease with central venous catheters

Exclusion Criteria:

* No central venous catheter
* Current CRBSI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing hemodialysis using a central venous catheter and Patients with underlying hematooncologic disease with central venous catheters
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2011-10; Primary Completion 2015-12 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
development of crbsi | Participants will be followed for the development of CRBSI during the duration of central venous catheter usage, an expected average of 1 year in hemodialysis patients and an expected average of six weeks in HSCT patients.
  There is only one outcome measure that is evaluated in two patient cohorts. Screening of catheter blood for microbial burden is performed during the whole study. Outcome measure is the development of CRBSI in these screened patients. Patients on hemodialysis using a CVC will be screened and observed for an sheduled time of approx. 1,5 years or until the CVC will be removed and hemodialysis no longer necessary. Patients undergoing HSCT will be screened and observed until CVC will be removed.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Krause, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz, Graz, Stmk, Austria